CLINICAL TRIAL: NCT04341779
Title: Simplifying Treatment and Monitoring for HIV (STREAM HIV): Point-of-Care Urine Tenofovir Adherence and Viral Load Testing to Improve HIV Outcomes in South Africa
Brief Title: Simplifying Treatment and Monitoring for HIV (STREAM HIV)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centre for the AIDS Programme of Research in South Africa (Network)
Responsible Party: Principal Investigator, Paul Drain, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00007544; R01AI147752 (NIH)
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: HIV/AIDS; HIV-1-infection
Keywords: Point-of-care test; Tenofovir; Adherence; HIV viral load
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Point-of-care adherence testing and Point-of-care viral load testing
  Interventions: Combination Product: Point-of-care viral load testing and tenofovir adherence testing
- Standard-of-care arm (No Intervention): No adherence testing and lab-based viral load testing

INTERVENTIONS:
Combination Product: Point-of-care viral load testing and tenofovir adherence testing — Point-of-care testing of HIV viral load and tenofovir, and providing same day results to participants
  Arms: Intervention arm

SUMMARY:
This study seeks to determine the clinical efficacy and cost effectiveness of implementing an integrated model for HIV monitoring using point of care (POC) tenofovir (TFV) adherence testing and POC viral load (VL) monitoring in improving ART adherence, maintaining durable VL suppression, and improving retention in care among HIV-positive individuals initiating first-line tenofovir disoproxil fumarate (TDF)-based ART in South Africa.

DETAILED DESCRIPTION:
This study will be a two-arm, open-label, randomized controlled superiority trial at an HIV clinic in Durban. HIV-positive individuals aged 16 years and above, who are initiating a tenofovir-based, first-line ART will be randomized to receive POC VL testing and POC TFV adherence testing, versus standard-of-care (SoC) viral load testing. The schedule for VL testing and management of VL test results will follow South African guidelines for HIV VL testing after ART initiation. 540 participants will be randomized (1:1) at ART initiation into the intervention arm (routine POC TFV adherence testing with POC VL monitoring) or the standard-of-care (SoC) arm (no objective TFV adherence testing and SoC VL monitoring).

Participants will be followed to compare concentrations between study arms at 24 weeks after ART initiation and a composite outcome of VL suppression and retention in care between the study arms at 72 weeks after ART initiation. The study will use process evaluation data, interviews and focus groups with patients and staff to assess implementation of the POC assays. Micro-costing will be conducted to estimate intervention costs.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* ≥16 years old
* Initiating a TDF-based, first-line ART regimen
* Do not self-report being on an ART regimen in the prior month
* Willing/able to provide written informed consent

Exclusion Criteria:

* Does not plan to continue receiving HIV care at the CDC Clinic
* Per the decision or opinion of the PI (for example, a clinically significant acute or chronic medical condition or circumstances that would make the patient unsuitable for participation or jeopardize the safety or rights of the participant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean tenofovir diphosphate concentration levels in dried blood spots | 24 weeks after ART initiation
  We will measure tenofovir-diphosphate concentrations in 3mm dried blood spots using liquid chromatography/tandem mass spectrometry.
Combined measure of virological suppression | 72 weeks after ART initiation
  We will measure viral load by a laboratory-based reference assay, performed by the South African National Health Laboratory Services. Viral suppression will be defined as a viral load <200 copies/mL.
Geometric mean TFV-DP concentrations similar among intervention and control participants | 24 weeks
  Participants with TFV-DP measured in the standard-of-care arm was 234, and in the intervention arm 242. With predetermined TFV-DP concentration thresholds for TFV-DP >200 flol/punch was 217 (92.7%) on the standard-ofcare arm and 239 (98.8%) on the Intervention arm. TFV-DP >750 fmol/punch was 199 (85.0%) and 210 (86.8%) with the intervention arm. However, predetermined analysis of TVF-DP thresholds showed more participants in the intervention arm achieved detectable TFV levels.
TFV-diphosphate (TVF-DP) concentrations in dried blood spots (DBS) as a long-term metric of adherence. | 24 weeks
  We will use Intracelllular TFV-DP concentrations (continuous) in DBS using liquid chromatography/tanem mass spectrometry at a certified lab.VL measured on stored samples across study arms using the Abbott Alinity assay--comparing continuaous log TFV-DP concentrations using t-tests and compared proportions with estimated risk rations (RR) using modified Poisson regression.

SECONDARY OUTCOMES:
Acceptability of point-of-care tenofovir and viral load testing | 24 and 72 weeks after ART initiation
  We will assess acceptability of point-of-care tenofovir and viral load testing by conducting semi-structured in-depth interviews and focus group discussions with study participants.
Cost-effectiveness of providing routine point-of-care tenofovir and viral load testing as compared to standard-of-care viral load monitoring | 24 and 72 weeks after ART initiation
  We will conduct a micro-costing of the costs associated with point-of-care tenofovir and viral load testing and will estimate the cost-effectiveness of the intervention using an existing individual-based, stochastic HIV model for KwaZulu-Natal for simulating health and economic outcomes.
Retention in care | 24 weeks
  This will be measured through attendance logs to assess ability to meet visit window goals.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Drain, MD, MPH, Principal Investigator — University of Washington; Nigel Garett, MBBS, PHD, Principal Investigator — Centre for the AIDS Programme of Research in South Africa (CAPRISA)
Locations (1):
- Centre for the AIDS Programme of Research in South Africa (CAPRISA), University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study will be made available
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following publication of primary results.
Access Criteria: De-identified data generated under this project will be administered in accordance with University of Washington, CAPRISA, and NIH policies, including the NIH Data Sharing Policy and Implementation Guidance of March 5, 2003.

REFERENCES:
- [Derived] Wang M, Moodley P, Khanyile M, Bulo E, Zondi M, Naidoo K, Sookrajh Y, Dorward J, Gandhi M, Garrett N, Drain PK, Sharma M. Cost and clinical flow of point-of-care urine tenofovir testing for treatment monitoring among people living with HIV initiating ART in South Africa. J Int AIDS Soc. 2025 Jul;28(7):e70004. doi: 10.1002/jia2.70004. PMID 40660747
- [Derived] Bardon AR, Dorward J, Sookrajh Y, Sayed F, Quame-Amaglo J, Pillay C, Feutz E, Ngobese H, Simoni JM, Sharma M, Cressey TR, Gandhi M, Lessells R, Moodley P, Naicker N, Naidoo K, Thomas K, Celum C, Abdool Karim S, Garrett N, Drain PK. Simplifying TREAtment and Monitoring for HIV (STREAM HIV): protocol for a randomised controlled trial of point-of-care urine tenofovir and viral load testing to improve HIV outcomes. BMJ Open. 2021 Oct 5;11(10):e050116. doi: 10.1136/bmjopen-2021-050116. PMID 34610939